CLINICAL TRIAL: NCT05163444
Title: Gait Analysis of Hemiparetics Adults Patients With Quadripod Cane and Rolling Cane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Maillard Berengere, Principal Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Liege Hospital Ethic Comittee
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Hemiplegic Gait
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic | interventions — Gait Analysis

STUDY DESIGN:
Intervention Model Description: Clinical trial, randomized, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rolling can (Experimental): Gait analysis with rolling cane
  Interventions: Device: Gait analysis with rolling cane
- Quadripod can (Active Comparator): Gait analysis with quadripod cane
  Interventions: Device: Gait analysis with quadripod cane

INTERVENTIONS:
Device: Gait analysis with rolling cane — 6 minutes walking test 10 meters walking test Before this experimentation, we will fix wearables sensors on the shoes.
  Arms: Rolling can
Device: Gait analysis with quadripod cane — 6 minutes walking test 10 meters walking test Before this experimentation, we will fix wearables sensors on the shoes.
  Arms: Quadripod can

SUMMARY:
After stroke, a lot of patients present an hemiparesis and gait disorders. They need walking aids like quadripod cane or rolling cane.

The quadripod cane confers a great stability but implies a walk in 3 times, thus consume more energy. The pause time necessary for the displacement (uplift) of the cane disappear with the Wheeleo.

The investigators will study many spatio-temporal parameters to determine which one allows to decrease the walking speed.

DETAILED DESCRIPTION:
Hemiparesis affects 65% of stroke patients and cause gait disorders. During rehabilitation, patients often need technical aids to the the return to walk.

For example, they can use the quadripod cane and the rolling cane, called Wheeleo. Regarding the first one, as its name indicate, there are 4 feet while the other model has 4 wheels.

Deltombe and al. proved that the walking speed is higher with a rolling cane. The investigators will recruited stroke patients and study many spatio-temporal parameters with a gait analysis system, when participants are walking with the two walking aids.

Participants will achieve 6 minutes walking test and a 10 meters walking test, with a wearable inertial systems on their shoes.

The investigators wish to reveal which spatio-temporal parameters most influence walking speed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Hemiparesis following a stroke
* Be able to walk with a quadripod cane independently
* Be able to walk with the rolling cane independently
* Be able to follow instructions

Exclusion Criteria:

* cognitive impairment
* acute orthopedic impairment
* other pathologies affecting walking (Parkinson's disease, severe polyneuropathy,...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-26 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
10 meters walking test at fast speed | 2 days
  Calculate the walking speed

SECONDARY OUTCOMES:
6 minutes walking test at spontaneous speed | 2 days
  Spatio-temporals factors analysis (symmetry, time of unipodal/bipodal stance station,...)

CONTACTS AND LOCATIONS:
Overall Officials: Berengere Maillard, Principal Investigator — University of Liege
Locations (2):
- Belgium (2):
  - CHUOA, Esneux, Liege
  - CNRF, Tinlot, Liege